CLINICAL TRIAL: NCT05215028
Title: Optimization of Mother-child Dyad Follow-up by a Multidomain Application: Real-world Cross Sectional Study
Acronym: MALO_2
Status: Completed | Type: Observational
Sponsor: Weprom (Other)
Collaborators: Kelindi (Industry)
Responsible Party: Sponsor
Other Study IDs: WP-2022-02
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Child Development Disorder; Post Partum Depression
MeSH Terms: conditions — Developmental Disabilities; Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- users: users of the web-application MALO
  Interventions: Device: web-application

INTERVENTIONS:
Device: web-application — web application multi-domain familial digital health record PRO The aim is to help for early screening of neurodevelopmental disorders of toddler after birth to 3 years of age and mother's postnatal depression, to improve vaccinations rate of toddlers and to provide advice to parents for child development.
  Other Names: MALO

SUMMARY:
After birth, the mother-child dyad can be impacted by issues which are usually under-detected or detected at early stage. Among these issues, neurodevelopmental disorders (NDD) such as autism spectrum disorder are common and affect 1 in 59 children but are detected after 4 years of age although it could be detected using parent report screens as early as 12 or 18 months of age. Moreover, parents are the main contributors of the screening of NDD in their children. In a recent French survey, the identification of the first symptoms was done by parents in 61% of cases and a health professional in only 14% and the mean age of disease detection was 6.8 years for autism spectrum disorder.

Other troubles that deserve early screening are hearing disorders which are observed in 1 child in 300 at 3 years of age and the main visual trouble in toddlers such as amblyopia which is observed with a prevalence of 3%.

Another issue that deserves improvement is the rate of mandatory or recommended vaccines in toddler which is only 71% for C-meningococcus and 79% for measles or rubella.

Concerning the mother, postnatal depression is defined as an episode of minor or major depression occurring during the first year postpartum with a pooled prevalence of 17.7%. Despite the high prevalence of this disorder and its potential impact on child development it remains underdetected and undertreated in daily practice.

The common point between all these disorders is that they can benefit from early detection by questionnaires intended for parents for their children or for themselves, because early treatment improves prognosis or prevent diseases.

An "all-in-one" multi-domain familial digital health record Patient reported outcomes application has been developing to help for early screening of neurodevelopmental disorders of toddler after birth to 3 years of age and mother's postnatal depression, to improve vaccinations rate of toddlers and to provide advice to parents for child development. The aim of the study is to assess in a real-world data-based the performances of this application.

ELIGIBILITY:
Inclusion Criteria:

* Parent of child or more under 3 years of age
* User of application Malo

Exclusion Criteria:

* Parent of a child who has already been diagnosed with a developmental disorder, known physical or mental disability

Max Age: 3 Years | Sex: All
Age Groups: Child
Study Population: The population includes all users of the Malo application, who did not object to the use of their data over the period from 11/11/2021 to 01/07/2022.
Sampling Method: Non-Probability Sample
Enrollment: 4346 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
impact on neurodevelopmental disorders detection | 3 years
  description of the rate and age at detection of each type of neurodevelopmental desorder
impact on hearing disorders | 3 years
  description of the rate and age at detection
impact on visual disorders | 3 years
  description of the rate and age at detection
impact on mandatory or recommended vaccines | 3 years
  rate of vaccines
impact on postnatal depression | 3 years
  rate of women in post natal depression

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice DENIS, Pr, Principal Investigator — ILC
Locations (1):
- ILC, Le Mans, France

IPD SHARING:
Plan to Share IPD: No